CLINICAL TRIAL: NCT01137695
Title: Symlin® Dose Escalation Efficacy vs. Conventional Therapy in Type 2 Diabetes Mellitus
Brief Title: Efficacy Study of High Dose Symlin to Treat Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cheryl Rosenfeld, DO (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor-Investigator, Cheryl Rosenfeld, DO, Principal Investigator, North Jersey Endocrine Consultants, LLC
Organization: North Jersey Endocrine Consultants, LLC (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEFCon2
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2011-10-14 (Estimated); Status verified 2011-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: pramlintide; glucose; type 2 diabetes mellitus; amylin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — pramlintide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Symlin Naive, Usual Dose (Active Comparator): Symlin 120 mcg three times daily in patients not previously treated with pramlintide before the study.
  Interventions: Drug: Pramlintide
- Symlin Naive, Dose Escalation (Experimental): Escalation of pramlintide dose to 360 mcg three times daily in patients not taking pramlintide prior to study.
  Interventions: Drug: Pramlintide
- Symlin treated, Usual Dose (Active Comparator): pramlintide 120 mcg three times daily in patients who have been treated with pramlintide 120 mcg prior to the trial.
  Interventions: Drug: Pramlintide
- Symlin Treated, Dose Escalation (Experimental): pramlintide 360 mcg three times daily in patients previously treated with 120 mcg prior to the study.
  Interventions: Drug: Pramlintide

INTERVENTIONS:
Drug: Pramlintide — 120 mcg SQ three times daily for 6 months.
  Arms: Symlin Naive, Usual Dose
Drug: Pramlintide — 360 mcg SQ three times daily for 6 months
  Arms: Symlin Naive, Dose Escalation
Drug: Pramlintide — 120 mcg SQ three times daily for 6 months
  Arms: Symlin treated, Usual Dose
Drug: Pramlintide — 360 mcg SQ three times daily for 6 months
  Arms: Symlin Treated, Dose Escalation

SUMMARY:
The hypothesis of the study is that those obese patients with type 2 diabetes mellitus who do not respond to the FDA approved dose of 120 mcg of pramlintide (Symlin®) 3 times daily with expected glucose control require higher than FDA approved dosage.

The primary objective of the study is to determine whether higher doses of pramlintide (Symlin®) in patients with type 2 diabetes mellitus control glucose better than the FDA approved dose of 120 mcg three times daily.

The secondary objectives include proving whether higher dose pramlintide (Symlin®) is more efficacious in causing weight loss and reduction in waist circumference than standard dose pramlintide (Symlin®),to determine whether blood levels of certain hormones correlate with need for higher dose therapy,and to determine whether or not the rate of common adverse effects exceeds the maximum FDA approved pramlintide (Symlin®) dose of 120 mcg three times daily.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years.
2. Type 2 diabetes mellitus.
3. Obese (BMI > 30 kg/m2), waist circ. >35" women, >40" men.
4. Basal insulin plus at least 2 injections of mealtime insulin daily or pre-mixed insulin.
5. On stable insulin dose for at least 3 mos (baseline + 20%, no minimum).
6. If pramlintide treated, on stable full dose for at least 3 months.
7. A1c > 7.0% and < 9.0%.
8. Women of childbearing age if using a reliable form of birth control.
9. Women of childbearing age if post tubal ligation or surgical menopause.
10. Able to consent.
11. Willing to perform self-monitoring of glucose.
12. Willing to attend study visits.
13. Written informed consent to participate in the study.
14. Agreement to maintain prior diet and exercise throughout the full course of the study.

Exclusion Criteria:

1. Age <18 or >80 years.
2. Confirmed gastroparesis or taking medications affecting gastric motility.
3. A1c <7.0% or >9.0%.
4. Recurrent severe hypoglycemia or hypoglycemic unawareness.
5. CHF.
6. Creatinine clearance <30 ml/min.
7. History of MI <6 mos prior to enrollment.
8. History of ventricular arrhythmia.
9. History of cancer or chemotherapy <6 mos prior to enrollment.
10. Laboratory abnormalities as follows:

    1. Liver enzymes >3X ULN.
    2. Hematocrit less than 30.
    3. Serum creatinine >2.5 mg/dl.
    4. Fasting triglycerides >500 mg/dl.
11. Cirrhosis.
12. Pregnancy or nursing.
13. Inability to provide consent.
14. Unwilling to attend study visits.
15. Unwilling to perform self-monitoring of glucose.
16. Chronic oral or parenteral glucocorticoid therapy (over one week of treatment) within 3 months prior to screening.
17. Investigational drug treatment within 3 months prior to screening.
18. Donation of blood, significant blood loss or transfusion within 3 months of screening.
19. History of acromegaly or Cushing's syndrome.
20. Use of prohibited concomitant medications.
21. Type 1 diabetes mellitus.
22. Acute metabolic complication (hyperosmolar state) <6 months prior to screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-01 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Glucose control | 6 months
  A1c Fasting plasma glucose Post-prandial glucose Glycomark

SECONDARY OUTCOMES:
Weight loss | 6 months
  Weight, BMI, Waist circumference.
amylin level | initial
  does initial blood amylin level correlate with need for higher dose pramlintide?
glucagon level | 6 months
  Does change in glucagon level correlate with glycemic response.
adverse effects | 6 months
  Whether or not the rate of common adverse effects exceeds the maximum FDA approved pramlintide (Symlin®) dose of 120 mcg TID (as compared to the clinical practice study) - GI: nausea 30% and Hypoglycemia: medically assisted 0.7% or patient ascertained 0.7%.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Rosenfeld, DO, Principal Investigator — North Jersey Endocrine Consultants; Jeffrey Rothman, MD, Principal Investigator — University Physicians Group Research; Alan Schorr, DO, Principal Investigator — St. Mary's Medical Center
Locations (3):
- United States (3):
  - North Jersey Endocrine Consultants, Denville, New Jersey
  - University Physicians Group, Staten Island, New York
  - St. Mary Medical Center, Langhorne, Pennsylvania